CLINICAL TRIAL: NCT00244478
Title: Influence of Soy on Bone Turnover and Body Composition in College Females
Brief Title: Soy, Bone and Health in College Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Dr. Richard D. Lewis, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-20-2005-FOCUS
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis; Obesity
MeSH Terms: conditions — Osteoporosis; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy Protein Dietary Supplement (Experimental): The soy-based meal replacements will contain 20 g soy protein and 161.2 mg isoflavones, 220-240 kcal, 31-36 g total carbohydrates, 0-2 g dietary fiber, 500 mg calcium, and 2.0-2.5 g total fat per serving.
  Interventions: Dietary Supplement: Soy Protein Dietary Supplement
- Placebo (Placebo Comparator): The control shake will have 20 g casein substituted for soy protein, and will be otherwise identical to the soy shakes. The shakes will be available in two flavors: chocolate and vanilla.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soy Protein Dietary Supplement — The soy-based meal replacements will contain 20 g soy protein and 161.2 mg isoflavones, 220-240 kcal, 31-36 g total carbohydrates, 0-2 g dietary fiber, 500 mg calcium, and 2.0-2.5 g total fat per serving.
  Arms: Soy Protein Dietary Supplement
Dietary Supplement: Placebo — The control shake will have 20 g casein substituted for soy protein, and will be otherwise identical to the soy shakes. The shakes will be available in two flavors: chocolate and vanilla.
  Arms: Placebo

SUMMARY:
This is a 16-week intervention to determine the efficacy of an isoflavone-rich soy based meal supplement to improve bone health and prevent weight and fat gain in 18-19 year old college females. The primary hypothesis is that participants who receive soy will have favorable changes in blood markers of bone and less weight and fat gain. The soy is provided by Physicians Pharmaceuticals, Inc. (Revival Doctor-formulated soy protein).

DETAILED DESCRIPTION:
The proposed study will be a 16-week randomized, double-blind, placebo-controlled trial designed to test whether a daily isoflavone-rich, soy-based meal replacement Revival Soy shake promotes favorables changes in bone biomarkers and attenuates weight gain in female college students. First-year college females were selected because of the potential for significant weight gain during their freshman year. The study will have a parallel design with two groups: the soy treatment group (SOY; n = 60) and a casein-based control (CON; n = 60). Exclusion criteria include significant weight loss or gain in the past 3 months, vegetarians and heavy soy food consumers, National Collegiate Athletic Association Division I athletes, women with eating disorders, present illnesses, chronic disease, and those taking medications or herbal supplements known to affect body weight, body fat or bone. Participants will be stratified based on BMI (18.0-24.9; 25-29.9; ≥30.0) and randomized to either SOY or CON groups.

Female college freshmen enrolled at the University of Georgia will be recruited in the fall of 2005. The soy-based meal replacements will contain 20 g soy protein and 161.2 mg isoflavones, 220-240 kcal, 31-36 g total carbohydrates, 0-2 g dietary fiber, 500 mg calcium, and 2.0-2.5 g total fat per serving. The control shake will have 20 g casein substituted for soy protein, and will be otherwise identical to the soy shakes. The shakes will be available in two flavors: chocolate and vanilla.

ELIGIBILITY:
Inclusion Criteria:

* 18-19 year old University of Georgia college females of all races/ethnicities.

Exclusion Criteria:

* significant weight loss or gain, currently dieting to lose weight, are planning to lose weight, diet or begin an exercise program, under the age of 18, pregnant or intending to become pregnant, vegetarians, heavy soy food consumers, Division I athletes, women with menstrual irregularities, eating disorders, present or chronic illness, and those taking medications known to affect bone, body weight or body fat.

Ages: 18 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bone specific alkaline phosphatase, N-telopeptide, osteocalcin, pyridinoline, deoxypyridinoline, height, weight, waist circumference, fat mass, fat-free soft tissue mass and bone mass will be measured at baseline, 8- and 16-weeks.

SECONDARY OUTCOMES:
Leptin, adipose tissue vascular endothelial growth factors, angiopoietins, and cytokines will be measured in the serum at baseline, 8- and 16-weeks. The impact of soy on satiety and depression will be measured at baseline, 8- and 16-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Lewis, Principal Investigator — The University of Georgia
Locations (1):
- The University of Georgia, Athens, Georgia, United States